CLINICAL TRIAL: NCT01849458
Title: BioFiber and BioFiber-CM Absorbable Biologic Scaffold for Soft Tissue Repair and Reinforcement Post-Market Surveillance Clinical Study
Brief Title: BioFiber Scaffold Post-Market Observational Study
Status: Completed | Type: Observational
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: Tornier 2013-1
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Results first posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Full Thickness Rotator Cuff Tear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BioFiber: Subjects implanted with BioFiber Scaffold or BioFiber-CM Scaffold
  Interventions: Device: BioFiber

INTERVENTIONS:
Device: BioFiber — Subjects implanted with BioFiber or BioFiber-CM Scaffold
  Other Names: BioFiber Scaffold; BioFiber-CM Scaffold

SUMMARY:
The aim of this study is to collect and report data from a consecutive series of patients implanted with these products as part of a post-market surveillance plan for CE Mark approval in the European Union.

DETAILED DESCRIPTION:
Rhe BioFiberTM Scaffold post-market surveillance study is a prospective, single arm, multi-center observational study with sites in the US and France.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older

  * Patients with full thickness rotator cuff tears (confirmed at time of surgery) that are eligible for rotator cuff repair.
  * Patients willing and able to comply with the requirements of the study protocol and provide informed consent.

Exclusion Criteria:

* Patients with active or latent infection
* Patients with decreased vascularity
* Patients with pathological soft tissue conditions
* Patients with a known allergy or sensitivity to tetracycline hydrochloride or kanamycin sulfate
* Patients with a known allergy or sensitivity to bovine collagen (BioFiber-CM only)
* Participating in a concurrent study that has not been approved for concurrent enrollment by the Clinical Study Manager

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orthopedic referral clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Brockmeier, MD, Principal Investigator — University of Virginia; Timothy Reish, MD, Principal Investigator — Insall Scott Kelly Institute; Philippe Collin, MD, Principal Investigator — St. Gregoire, France
Locations (3):
- United States (2):
  - Insall Scott Kelly Institute, New York, New York
  - University of Virginia Sports Medicine and Shoulder Surgery, Charlottesville, Virginia
- St. Gregoire, Saint-Grégoire, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Single arm
Groups:
- BioFiber Scaffold: Single arm of subjects implanted with BioFiber Scaffold or BioFiber-CM Scaffold
Period: Overall Study
Arm/Group | BioFiber Scaffold
Started | 50; 50 Single arm
6 Months Follow-up | 50; 50 Single arm
Completed | 46; 46 Single arm
Not Completed | 4; 4 Single arm
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Units Other Than Participants: Arms
Arm/Group | BioFiber
Number analyzed (Participants) | 50
Number analyzed (Arms) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 39
  France | 11
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.9 (7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Device Associated Adverse Events
Description: The primary objective is to report the number of participants with device associated adverse events.
  Device associated adverse events are defined as adverse events that are classified as possibly or definitely related to the study product or procedure, or anticipated adverse events listed in the product's Instruction for Use regardless of relationship to the study device.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | BioFiber
Number analyzed (Participants) | 46
Participants | 4

2. Secondary Outcome: Clinical Functional Outcome - Adjusted Constant-Murley Score
Description: Evaluate clinical functional outcome Adjusted Constant-Murley Score. The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient.[1] The Constant-Murley score was introduced to determine the functionality after the treatment of a shoulder injury. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher the score, the higher the quality of the function. A score of 0 is considered the worst outcome and 100 is considered the best outcome.
Time Frame: 6 Months
Population: 50 Participants
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BioFiber
Number analyzed (Participants) | 50
scores on a scale | 93.4 (17.5)
Statistical Analysis 1: Comparison: BioFiber; Difference from baseline (6M-Baseline); Test type: Superiority or Other; p = 0.0001, 2-sided, paired t-test; Mean Difference (Final Values) = 32.6, 95% CI 2-sided [25.2 to 40], Standard Deviation 26

3. Secondary Outcome: Clinical Functional Outcome - Adjusted Constant-Murley Score
Description: as for outcome 2
Time Frame: 12 Month
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BioFiber
Number analyzed (Participants) | 46
scores on a scale | 97.1 (16.1)
Statistical Analysis 1: Comparison: BioFiber; Difference from baseline (12M-Baseline); Test type: Superiority or Other; p = 0.0001, 2-sided, paired t-test; Mean Difference (Final Values) = 35.7, 95% CI 2-sided [28.7 to 42.7], Standard Deviation 23.6

4. Secondary Outcome: Clinical Functional Outcome - WORC Index
Description: Evaluate clinical functional outcome WORC Index. This is a quality-of-life measurement specific for rotator cuff disease based on 21 questions answered using visual analog scales. It is organized in 5 subscales: physical symptoms, sprots/recreation, work, lifestyle, and emotions. Each item has a possible score from 0-100 where higher scores represent a lower quality of life. The scores are summed up to a possible 2100 points. The total number of points is subtracted from 2100, divided by 2100, then multiplied by 100 to create a percentage. The final score is thus a percentage ranging from 0 to 100 with higher percentages indicating better quality of life.
Time Frame: 6 Months
Population: One subject is missing data for this outcome measure thus a total of 49 subjects were analyzed in this section.
Measure: Mean (Standard Deviation); unit: Percentage of WORC Index
Arm/Group | BioFiber
Number analyzed (Participants) | 49
Percentage of WORC Index | 80.7 (18.9)
Statistical Analysis 1: Comparison: BioFiber; Difference from baseline (6M-Baseline); Test type: Superiority or Other; p = 0.0001, 2-sided, paired t-test; Mean Difference (Final Values) = 43.8, 95% CI 2-sided [37.4 to 50.1], Standard Deviation 22.2

5. Secondary Outcome: Clinical Functional Outcome - WORC Index
Description: as for outcome 4
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: Percentage of WORC Index
Arm/Group | BioFiber
Number analyzed (Participants) | 46
Percentage of WORC Index | 86.8 (16.3)
Statistical Analysis 1: Comparison: BioFiber; Difference from baseline (12M-Baseline); Test type: Superiority or Other; p = 0.0001, 2-sided, paired t-test; Mean Difference (Final Values) = 49.2, 95% CI 2-sided [43.2 to 55.2], Standard Deviation 20.2

6. Secondary Outcome: Number of Study Participants With Re-tears
Description: Assess re-tears of the repaired tendon using ultrasound imaging. The definition of a re-tear for the rate reported is any full thickness tear in a tendon that was repaired with the BioFiber Scaffold that is at least 80% of the size of the original tear.
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | BioFiber
Number analyzed (Participants) | 50
Participants | 2

7. Secondary Outcome: Number of Study Participants With Re-tears
Description: as for outcome 6
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | BioFiber
Number analyzed (Participants) | 46
Participants | 2

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | BioFiber
Serious Adverse Events (participants affected / at risk) | 3/50
Other Adverse Events (participants affected / at risk) | 1/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BioFiber (N=50)
Infection (Infections and infestations) | 1 (1) — Left shoulder deep abscess and suspected septic arthritis of glenohumeral joint. Not related to device, possible relatedness to procedure.
Stroke (Vascular disorders) | 1 (1) — Acute ischemic Stroke, multiple punctate infarcts in the first posterior, frontal and parietal lobes. Not related to device, not related to procedure.
Deep Vein Thrombosis (Vascular disorders) | 1 (1) — Deep Vein Thrombosis/pulmonary embolism. Not related to device, possible relatedness to procedure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BioFiber (N=50)
Clot (Vascular disorders) | 1 (1) — Focal 1 cm superficial clot in mid left basilica vein. Reported as not related to device and possibly related to procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No